CLINICAL TRIAL: NCT07270159
Title: EFFECT OF PROBIOTICS, DOUBLE ANTIBIOTIC AND CALCIUM HYDROXIDE PASTE AS INTRACANAL MEDICAMENTS ON POSTOPERATIVE PAIN IN SYMPTOMATIC IRREVERSIBLE PULPITIS PATIENTS. A RANDOMIZED CONTROLLED TRIAL
Brief Title: Effect of Probiotics, Double Antibiotic Paste, and Calcium Hydroxide on Postoperative Pain in Irreversible Pulpitis: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Zainab Dua, Lecturer, Dow University of Health Sciences
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 181
Record Dates: First submitted 2025-11-24; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-05

CONDITIONS: Root Canal Treatment; Irreversible Pulpitis With Apical Periodontitis; Pulpitis - Irreversible; Post Operative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcium Hydroxide (Active Comparator): Intrcanal medicament used in RCT
  Interventions: Drug: Probiotic
- Double Antibiotic Paste (DAP) (Active Comparator): Intracanal medicament used in RCT
  Interventions: Drug: Probiotic

INTERVENTIONS:
Drug: Probiotic — New intracanal medicament used in RCT

SUMMARY:
The goal of this clinical trial is to learn whether probiotics, double antibiotic paste (DAP), or calcium hydroxide paste help reduce postoperative pain after root canal treatment in adults with symptomatic irreversible pulpitis.

It will also learn about the safety of these medicaments.

The main questions it aims to answer are:

Do probiotics, DAP, or calcium hydroxide lower the amount of pain patients experience after the first visit of root canal treatment? What medical problems or side effects do participants experience when any of these medicaments are used? Researchers will compare probiotics, DAP, and calcium hydroxide to see which one works best to control postoperative pain.

Participants will:

Receive one of the three intracanal medicaments (probiotics, DAP, or Ca(OH)₂) placed inside their root canal Visit the clinic for follow-ups according to the treatment plan Report their pain levels using a Visual Analog Scale (VAS) at several time points (before treatment, 12 hrs, 24 hrs, 48 hrs, 3 days, and 7 days) Inform the research team about any discomfort, symptoms, or side effects during the week after treatment

DETAILED DESCRIPTION:
This randomized controlled clinical trial aims to evaluate the effectiveness of three intracanal medicaments-probiotics, double antibiotic paste (DAP), and calcium hydroxide-in reducing postoperative pain in adult patients diagnosed with symptomatic irreversible pulpitis undergoing root canal treatment. The study will compare changes in pain intensity over time using the Visual Analog Scale (VAS) and assess any adverse effects associated with each medicament. A total of 75 participants will be randomly assigned to one of the three treatment groups. The study seeks to determine which medicament provides the greatest reduction in postoperative pain and whether probiotics may serve as a safe and effective alternative to commonly used intracanal materials.

Detailed Description Postoperative pain following root canal treatment remains a significant clinical concern, particularly among patients with symptomatic irreversible pulpitis. Although calcium hydroxide is the most widely used intracanal medicament, its limitations-including delayed onset of action, high solubility, and limited antibacterial effectiveness against certain microorganisms-have led to increasing interest in alternative options. Double antibiotic paste, containing metronidazole and ciprofloxacin, has shown strong antimicrobial activity, while probiotics have recently emerged as a potential biotherapeutic alternative with antibacterial and anti-inflammatory properties.

This randomized controlled trial will compare the pain-reducing effectiveness of three intracanal medicaments: calcium hydroxide paste, double antibiotic paste, and a probiotic paste consisting of Lactobacillus rhamnosus GG. Participants aged 18-45 years who are diagnosed with symptomatic irreversible pulpitis, with or without symptomatic apical periodontitis, will be enrolled. After standardized root canal preparation, one of the three medicaments will be placed inside the canal during the first appointment.

Pain will be assessed using a 10-point Visual Analog Scale (VAS) at the following intervals:

Preoperative 12 hours postoperative 24 hours 48 hours 3 days 7 days Any adverse events or additional symptoms-such as swelling, fever, or severe recurrent pain-will be documented. Participants may use prescribed analgesics only if necessary. The medicament will be removed at the second visit after one week, followed by completion of root canal filling.

The study will include 75 participants, allowing for potential dropout, with 25 participants per treatment group. Randomization will be computer-generated, and the trial will be double-blinded, ensuring that neither the participants nor the outcome assessors are aware of group allocations.

The primary outcome is the change in postoperative pain intensity over time. Secondary outcomes include the incidence of adverse reactions and any differences in analgesic use among the three groups.

This study will provide valuable evidence to guide the selection of intracanal medicaments, assess the potential benefits of probiotics in endodontic pain management, and support the development of safer and more effective treatment strategies for patients with symptomatic irreversible pulpitis

ELIGIBILITY:
Inclusion Criteria:

1. Patients falling in ASA 1 category
2. Suffering from symptomatic irreversible pulpitis with range from moderate to severe. In addition to this patient should also have experienced lingering of pain. VAS score will be used to record pain. (Confirmed by clinical and radiographic signs) with or without apical periodontitis.
3. Multirooted teeth (Mandibular 1st and 2nd molars)
4. Age 18-45 year
5. Teeth with a Periapical Index (PAI) score of 1 -3, indicating a healthy periapical status or minimal changes in bone structure not necessarily associated with apical periodontitis, were included in this study.

Exclusion Criteria:

1. Pregnant or lactating mothers
2. Subjects taking chronic pain medications within last 24 hrs.
3. Cracks, complex anatomy, pulp calcification

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Intensity | Preoperative 12 hours postoperative 24 hours postoperative 48 hours postoperative 3 days postoperative 7 days postoperative
  Change in postoperative pain levels following root canal treatment, measured using the Visual Analog Scale (VAS). VAS is a 10-point scale where 0 = no pain and 10 = worst possible pain. Participants will report their pain at multiple time points to evaluate how each intracanal medicament (Calcium Hydroxide, Double Antibiotic Paste, Probiotic Paste) influences pain reduction over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Dow International Dental College, Karachi, Sindh, Pakistan